CLINICAL TRIAL: NCT06946706
Title: Assessing the Prevalence and Epidemiological Characteristics of Small Intestinal Bacterial Overgrowth (SIBO) in Patients With Autoimmune Gastritis (AIG) Through Hydrogen and Methane Breath Testing (HMBT).
Brief Title: Assessing the Prevalence and Epidemiological Characteristics of Small Intestinal Bacterial Overgrowth (SIBO) in Patients With Autoimmune Gastritis(AIG) Through Hydrogen and Methane Breath Testing(HMBT).
Acronym: HMBT、SIBO、AIG
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LY2024-318-A
Record Dates: First submitted 2025-04-19; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Autoimmune Gastritis
Keywords: small intestinal bacterial overgrowth(SIBO); hydrogen and methane breath testing(HMBT)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- the AIG group: Patients diagnosed with AIG: Previous gastroscopy (or) histological findings consistent with AIG, and serological tests support the diagnosis of AIG
  Interventions: Diagnostic Test: hydrogen and methane breath testing
- the acid suppression group: Patients who are non-AIG and need long-term acid inhibitor (PPI more than 8 weeks or P-CAB more than 4 weeks) due to gastroesophageal reflux and other reasons
  Interventions: Diagnostic Test: hydrogen and methane breath testing
- the control group: Patients with a 1-year history of gastroscopy, with no degree of microscopic atrophy, or with mild gastric mucosal atrophy (C-I and C-II according to the Kimura-Takemoto classification) and at least 2 weeks without taking PPI/P-CAB
  Interventions: Diagnostic Test: hydrogen and methane breath testing

INTERVENTIONS:
Diagnostic Test: hydrogen and methane breath testing — The hydrogen and methane breath testingt(HMBT) is a non-invasive method based on gas analysis of gut microbiota metabolomics.Normal human metabolic processes do not produce methane and hydrogen, and all methane and hydrogen in exhaled breath come from metabolites produced during the fermentation of substrates by gut microbiota. About 14-21% of the gas can diffuse through the intestinal mucosa to the bloodstream, circulate through the bloodstream to the alveoli, and be exhaled through gas exchange.Based on substrate properties, separate and measure methane and hydrogen concentrations from exhaled breath for non-invasive, convenient, and accurate diagnosis of microbial imbalance/small intestine bacterial overgrowth (SIBO)

SUMMARY:
Evaluate the prevalence of small intestinal bacterial overgrowth in patients with autoimmune gastritis (AIG) through hydrogen and methane breath testing, and determine whether there are differences in the positive rates of hydrogen and methane breath testing among the AIG group, the acid suppression group, and the control group.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the AIG group:

  1. Age range: 18-65 years old, without gender limitation;
  2. Patients diagnosed with AIG: Previous gastroscopy (or) histological findings consistent with AIG, and serological tests support the diagnosis of AIG;
  3. Previous colonoscopy or intestinal CT have ruled out inflammatory bowel disease, malignant tumors, history of pseudo and mechanical bowel obstruction, and there is currently no evidence to support these diseases;
  4. At least 2 weeks without taking PPI/P-CAB;
  5. Possessing the ability to independently or with the assistance of medical staff, complete hydrogen and methane breath tests and related questionnaire scoring;
  6. Capable of completing the signing of informed consent forms as required.

Inclusion criteria for the acid suppression group:

1. Age: 18-65 years old, without gender limitation;
2. Patients who are non-AIG and need long-term acid inhibitor (PPI more than 8 weeks or P-CAB more than 4 weeks) due to gastroesophageal reflux and other reasons;
3. Patients with a 1-year history of gastroscopy, with no degree of microscopic atrophy, or with mild gastric mucosal atrophy (C-I and C-II according to the Kimura-Takemoto classification);
4. Previous colonoscopy or intestinal CT have ruled out inflammatory bowel disease, malignant tumors, history of pseudo and mechanical bowel obstruction, and there is currently no evidence to support these diseases;
5. Possessing the ability to independently or with the assistance of medical staff, complete hydrogen and methane breath tests and related questionnaire scoring;
6. Capable of completing the signing of informed consent forms as required.

Inclusion criteria for the control group:

1. Age: 18-65 years old, without gender limitation;
2. Patients with a 1-year history of gastroscopy, with no degree of microscopic atrophy, or with mild gastric mucosal atrophy (C-I and C-II according to the Kimura-Takemoto classification);

4) Previous colonoscopy or intestinal CT have ruled out inflammatory bowel disease, malignant tumors, history of pseudo and mechanical bowel obstruction, and there is currently no evidence to support these diseases; 4) At least 2 weeks without taking PPI/P-CAB; 5) Possessing the ability to independently or with the assistance of medical staff, complete hydrogen and methane breath tests and related questionnaire scoring; 6) Capable of completing the signing of informed consent forms as required.

Exclusion Criteria:

* 1)Gastrointestinal endoscopy suggests patients with active gastrointestinal ulcers; 2)History of malignant tumors of the digestive system (not limited to the digestive tract), inflammatory bowel disease, and pseudo or mechanical bowel obstruction in the past; 3)Previous gastrointestinal resection surgery;appendectomy and cholecystectomy within 1 year; 4)History of gastrointestinal perforation, gastrointestinal bleeding, cholangitis, and acute or chronic pancreatitis within one year; 5)Evidence suggests current gastrointestinal infections (Helicobacter pylori, acute infectious enteritis); 6)History of type I diabetes and primary hypothyroidism (the patients with normal thyroid function can be included); 7)Diagnosed lactose malabsorption, lactose intolerance, and pancreatic exocrine dysfunction; 8)History of antibiotic use within four weeks; 9)History of endoscopic examination within two weeks; 10)History of taking gastrointestinal motility promoting drugs, probiotics, and laxatives within one week; 11)On the day before the test, consume fermentable foods such as yogurt, kimchi, soy sauce, oats, beer, etc; 12)Eight hours prior to testing, without fasting; 13)Smoking and vigorous exercise two hours before and during the testing period; 14)Difficulty in exhaling due to respiratory system diseases, or inability to fast or drink for extended periods of time, resulting in inability to complete hydrogen and methane breath tests; 15)Pregnant, lactating women, or those with poor overall compliance, or other situations that researchers consider necessary to exclude.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Chinese people
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
hydrogen and methane breath testing | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Institute of Digestive Disease, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No